CLINICAL TRIAL: NCT02005094
Title: The Role of Inflammasome in Inflammatory Macrophage in Mycobacterium Avium Complex-lung Disease and Mycobacterium Abscessus-lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201308008RINA
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: To Investigate the Inflammasome Response of Inflammatory and Resting Macrophage; To Compare the Difference of Inflammasome Response of Inflammatory Macrophage; To Study the Diagnostic Aid From Immunological Markers in Inflammasome Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy group: patients without MAC/MAB lung disease and colonization
- MAC/MAB colonization group: patients with pulmonary MAC/MAB colonization
- MAC/MAB lung disease group: Patient with MAC/MAB lung disease

SUMMARY:
1. To investigate the inflammasome response of inflammatory and resting macrophage derived from healthy human participants by stimulation using MAC or MAB bacilli.
2. To compare the difference of inflammasome response of inflammatory macrophage by MAC/MAB bacilli stimulation between MAC/MAB-LD patients and the colonizers.
3. To study the diagnostic aid from immunological markers in inflammasome response in inflammatory macrophage stimulated by MAC/MAB.

DETAILED DESCRIPTION:
Lung disease (LD) due to nontuberculous mycobacteria (NTM) becomes an important clinical concern, because the incidence and prevalence of NTM-LD have increased over the last decade. Among the NTM-LD in Taiwan, Mycobacterium avium complex (MAC) and M. abscessus (MAB) are the most frequent pathogenic species. Because MAC and MAB exist in the environment ubiquitously, clinical relevance of MAC isolated in sputum is only around 35~42%, and that of MAB is around 33%. According to the guideline of the American Thoracic Society, the diagnosis of MAC-LD and MAB-LD is based on clinical, radiographic, and mycobacteriologic criteria. For microbiology criteria, two or more sets of positive sputum mycobacterial culture for the same NTM species within one year is required. Actually, mycobacteria culture is neither timely nor efficient, which needs weeks to wait the results, especially for the slowly growing NTM. Moreover, the nucleic acid amplification method cannot discriminate true NTM infection and solely colonization because airway NTM colonization is not uncommon. Therefore, diagnosis of true NTM-LD is a big challenge in clinical practice. However, to early diagnose and then start treatment of NTM-LD is important because NTM-LD may be rapid lethal in critical status or in patients without early proper treatment. Hence, more rapid and accurate diagnostic test should be developed.

The body inflammatory markers are probably indicators for differentiating true NTM-LD from pulmonary colonization and interferon-gamma (IFN-g) play a critical role in protective immunity to mycobacterial infections. However, serum IFN-g poorly correlated with diagnosis of NTM-LD and possibly due to the hosts with attenuated cellular immunity and the presence of IFN-gamma inhibitor. By contrast, macrophages are the first-line defense while mycobacterial bacilli enter through airway and may play an important role while MAC/MAB infection. Macrophages can be polarized to inflammatory type and promotes type 1 immunity. In addition, inflammatory macrophages can react through inflammasome to defense intracellular mycobacteria. However, the inflammasome responses in inflammatory macrophages are rarely investigated in MAC-LD and MAB-LD, either for the defense mechanism or its diagnostic aid for disease form colonization. The investigators therefore conduct an in-vitro inflammatory macrophage stimulation using MAC or MAB bacilli to observe the difference of inflammasome response between MAC/MAB patients, colonizers, and controls.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* MAC/MAB lung disease: Diagnosis is based on the guidelines made by American Thoracic Society (Table 1)[1]. In brief, there should be pulmonary symptoms, comparable findings in chest image and appropriate exclusion other possible causes as well as meeting the microbiology criteria.
* MAC/MAB pulmonary colonizers: Those without fulfilling the diagnostic criteria but having at least one set of positive sputum for MAC/MAB are defined.
* Healthy controls: patient without documented MAC/MAB lung disease and pulmonary colonization

Exclusion Criteria:

* Patients who have acquired immunodeficiency syndrome
* Patients who have bleeding tendency which cannot tolerate venous puncture such as hemophilia, thrombocytopenia.
* refusal of recruitment

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥ 20 years
  2. MAC/MAB lung disease: Diagnosis is based on the guidelines made by American Thoracic Society (Table 1)[1]. In brief, there should be pulmonary symptoms, comparable findings in chest image and appropriate exclusion other possible causes as well as meeting the microbiology criteria.
  3. MAC/MAB pulmonary colonizers: Those without fulfilling the diagnostic criteria but having at least one set of positive sputum for MAC/MAB are defined.
  4. Healthy controls: patient without documented MAC/MAB lung disease and pulmonary colonization
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
survival | one year

SECONDARY OUTCOMES:
the amount of cytokine released by inflammatory macrophage | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan